CLINICAL TRIAL: NCT06361095
Title: Confirmatory Efficacy Trial of a Traditional vs. Gamified Attention Bias Modification for Depression
Brief Title: Confirmatory Efficacy Trial of Attention Bias Modification for Depression
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Arcade Therapeutics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01GABM
Record Dates: First submitted 2024-04-01; First posted 2024-04-11 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-05

CONDITIONS: Depression
Keywords: depression treatment; attention bias modification; digital mental health treatment
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sham Attention Bias Modification (Sham Comparator): Sham and traditional ABM interventions will be identical in all respects with one critical exception. For sham ABM, after stimuli offset the target will appear with equal probability (50%) in the location of the neutral or the dysphoric stimulus.
  Interventions: Behavioral: Sham Attention Bias Modification
- Traditional Attention Bias Modification (Active Comparator): This ABM variant is a web-based program delivered to participants via a computer. It presents pairs of stimuli to the right and left visual fields from two stimulus categories: sad or neutral facial expressions from the Pictures of Facial Affect (POFA) collection and dysphoric or neutral scenes from or from the International Affective Picture System (IAPS) collection.
  Interventions: Behavioral: Traditional Attention Bias Modification
- Gamified Attention Bias Modification (Experimental): This ABM variant will be completed on participants' mobile devices (iOS or Android). During app use, they will be presented with sad-happy stimulus pairs followed by target probes (tracing a path) always appearing at the happy stimulus location.
  Interventions: Behavioral: Gamified Attention Bias Modification

INTERVENTIONS:
Behavioral: Traditional Attention Bias Modification — Each ABM trial begins with a central fixation cross for 1500ms, followed by a pair of POFA or IAPS stimuli (see Figure 3). POFA pairs will be presented for 3000ms, while IAPS pairs will be presented for 4500ms (due to the increased image complexity of IAPS images relative to POFA images). Longer stimulus duration times were selected based on evidence that attention biases for sad stimuli are prolonged in depression. Following offset of the images, either a single or double asterisk probe appears in the location of one of the images and will remain until a participant response or 10,000ms. In active ABM, the probe had an 80% probability of appearing in the location of the neutral stimulus. Investigators selected 80% rather than 100% to allow for computing attention bias during training and to facilitate task engagement. At the end of each ABM session, participants are provided feedback regarding their task performance relative to their last five sessions in a visual format.
  Arms: Traditional Attention Bias Modification
Behavioral: Gamified Attention Bias Modification — Each trial consists of the fixation stage, facial cue stage, and response stage. At the fixation stage, an image appears (a colorful medallion) for 500 ms. The fixation appears randomly within a fixed rectangular field on the user's smartphone screen, and is always at the midpoint between the two face cues that will appear in the next stage. Next, after the cue disappears, two animated faces appear on the screen, one happy and one sad, with a 1000ms duration. Immediately after they disappear, a target probe (a trail) appears in the location of the happy face cue. The path remains (up to 3 seconds) until participants respond by tracing it starting from the point at which the face cue disappeared. They are instructed to quickly but accurately trace the path with their finger and receive visual and haptic feedback during tracing to indicate they are tracing accurately, followed by the path disappearing.
  Arms: Gamified Attention Bias Modification
Behavioral: Sham Attention Bias Modification — Sham attention bias modification designed to match the active ABM condition in all respects except for the shifting attention away from negative stimuli in active attention bias modification.
  Arms: Sham Attention Bias Modification

SUMMARY:
The goal of this clinical trial is to compare the efficacy of two related, but different ABM (Attention Biased Modification) treatments for depression in adults with elevated symptoms of depression. The main aims are:

* Aim 1:examine whether gamified ABM leads to greater change in the primary and secondary outcomes than sham ABM
* Aim 1: establish that gamified ABM is at least as effective as traditional ABM.
* Aim 2: identify moderators of ABM efficacy and mechanisms responsible for its efficacy.
* Aim 3: Identify the durability of ABM on depression symptoms during short-term follow-up

Participants will complete self-report questionnaires, complete eye-tracking tasks, and be clinically assessed through interviews by clinician researchers.

If there is a comparison group: Researchers will compare sham, traditional, and gamified treatment groups to see if they moderate symptoms of depression.

DETAILED DESCRIPTION:
The overall goal of this project is to conduct a well-powered confirmatory efficacy trial comparing a gamified, attention bias modification (ABM) mobile application and traditional ABM to sham ABM among adults with elevated symptoms of depression. The proposed R01 efficacy trial follows the NIMH intervention development sequence as it builds upon prior NIMH-funded experimental therapeutics work, specifically R21MH092430 "Attention training for Major Depressive Disorder" and R33MH109600 "Development of attention bias modification for depression". This prior work demonstrates that active ABM engages and alters negative attention bias and there is a preliminary efficacy signal that ABM reduces depression. Although traditional ABM is efficacious for the treatment of depression, "gamified" forms of ABM have the potential to be more accessible and engaging than traditional ABM. Pilot work suggests that a gamified ABM can reduce negative affect; however, its effectiveness for depression has not yet been established. Thus, investigators are proposing to conduct a well-powered, confirmatory efficacy trial to determine ABM's potential for the treatment of depression. In Aim 1, the investigators will examine the efficacy of ABM in a large sample of adults (N = 600) with elevated symptoms of depression. The investigators hypothesize that gamified and traditional ABM will lead to significantly greater reductions in self-reported and interviewer-rated depression symptoms than sham ABM. The investigators further hypothesize that traditional ABM will be non-inferior to gamified ABM (treatment superiority between the ABM conditions will also be tested). In Aim 2, the investigators will examine putative moderators and mediators of ABM. Based on ABM research with anxious populations, it is predicted that people with a strong initial attentional bias for sad stimuli will experience greater reductions in depression in response to either gamified or traditional ABM than sham ABM. In terms of mediation, compared to sham ABM, the investigators hypothesize that gamified and traditional ABM will: (1) decrease negative attentional bias measured behaviorally with reliable eye tracking methods; (2) significantly reduce depression; and (3) improve depression symptoms via their influence on negative attentional bias. Selection of the putative mediators is informed by our prior R33 ABM trial, where it was found that gaze bias away from sad stimuli mediated the effect of traditional ABM on depression symptom change. In Aim 3, an exploratory aim, the investigators will estimate the durability of ABM by collecting post-treatment symptom data 1-, 2-, 3-, and 6-months after ABM completion. Symptom change and reliable recovery across a six-month follow-up period will be estimated. Currently, the durability of ABM effects for depression is unknown, as few well-powered ABM studies for depression have obtained follow-up data. This trial would provide the most definitive data to date regarding whether ABM for depression is a promising treatment for depression.

ELIGIBILITY:
Inclusion Criteria:

* Provided informed consent
* Fluent in English
* Scored 13 or greater on the QIDS-SR at the baseline assessment
* Between the ages of 18 to 70
* Have had no changes in medication and dosage in the past 12 weeks (if currently on antidepressant medication)

Exclusion Criteria:

* Reported suicidal behavior or significant suicidal ideation within the past six months using the Columbia-Suicide Severity Rating Scale (C-SSRS)
* Met criteria for current or past bipolar or psychotic disorders
* Current (i.e., within the past 12 months) substance use disorders of moderate or greater severity on the Mini International Neuropsychiatric Interview (MINI)
* Currently taking opioid analgesics or systemic corticosteroid use as these medications
* Currently receiving psychotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
QIDS (Quick Inventory of Depression Symptoms) SR-16 | Screening, Baseline, Weeks 1-4 (Acute Period), Weeks 12-28 (Follow-Up Period)
  The Quick Inventory of Depressive Symptoms (QIDS) is a 16-item measure (self-report and clinician-rated versions) for adults with depression with solid psychometric properties and substantial data supporting sensitivity to change. The QIDS assesses the criterion domains used to diagnose a major depressive disorder.
  The participant must score a minimum of 13 on the QIDS-SR at the baseline assessment to qualify for participation. Total QIDS scores range from 0 to 27, with higher scores reflecting greater severity of depression, and thus, worst outcomes for our study.

SECONDARY OUTCOMES:
Sheehan Disability Scale (SDS) | Baseline, Weeks 1-4 (Acute Period), Weeks 12-28 (Follow-Up Period)
  Self-report measure of symptom-related disability. SDS total score ranges from 0 (unimpaired) to 30 (highly impaired). Higher scores mean a worse outcome.
Snaith-Hamilton Pleasure Scale (SHAPS) | Baseline, Weeks 1-4 (Acute Period), Weeks 12-28 (Follow-Up Period)
  Self-report measure of anhedonia severity. SHAPS total score ranges from 0 to 14, with higher scores meaning worse outcomes.
Hamilton Depression Rating Scale (HAM-D) | Baseline, Weeks 1-4 (Acute Period), Weeks 12-28 (Follow-Up Period)
  Interviewer-rated measure of depression symptom severity. Scoring for this assessment can range from a minimum total score of 0 (least severe) and a maximum score of 52 (most severe). Higher scores mean worse outcomes.
Generalized Anxiety Disorder (GAD-7) | Baseline, Weeks 1-4 (Acute Period), Weeks 12-28 (Follow-Up Period)
  Self-report measure of anxiety symptom severity. GAD-7 total score for the seven items ranges from 0 to 21, with higher scores indicating worse outcomes.
Perseverative Thinking Questionnaire (PTQ) | Baseline, Weeks 1-4 (Acute Period), Weeks 12-28 (Follow-Up Period)
  A content-independent measures of repetitive negative thinking. PTQ total score for 15 items ranges from 0 to 60, with higher scores indicating worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher G Beevers, PhD, Principal Investigator — UT Austin
Locations (1):
- Institute for Mental Health Research, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators will share data via the NDAR and code via the Texas Data Repository (https://dataverse.tdl.org/dataverse/mdl). The data is expected to become available at the end of the trial (~ 5 years from now). Qualified researchers, as determined by the NIH's NDAR, will have access to the data. Anyone can access the code. The Study Protocol will be shared via a publication in a protocol journal within the next year.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data is expected to become available at the end of the clinical trial (approximately five years from now) with no end date.
Access Criteria: Qualified researchers, as determined by the NIH's NDAR, will have access to the data.

REFERENCES:
- [Derived] Fadrigon B, Tseng A, Weisenburger RL, Levihn-Coon A, McNamara ME, Shumake J, Smits JAJ, Dennis-Tiwary TA, Beevers CG. Efficacy of traditional and gamified attention bias modification for depression: Study protocol for a randomized controlled trial. Contemp Clin Trials. 2025 Feb;149:107797. doi: 10.1016/j.cct.2024.107797. Epub 2024 Dec 24. PMID 39725004

DOCUMENTS (1):
  • Informed Consent Form (2024-04-05): https://cdn.clinicaltrials.gov/large-docs/95/NCT06361095/ICF_000.pdf